CLINICAL TRIAL: NCT05420688
Title: The Turkish Validity-Reliability Study of the European Heart Failure Self-Care Behavior Scale-Caregivers Version (AKYÖDÖ-BV)
Brief Title: The Turkish Validity-Reliability Study of the European Heart Failure Self-Care Behavior Scale-Caregivers Version
Status: Completed | Type: Observational
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, İbrahim Caner Di̇ki̇ci̇, Lecturer, Harran University
Other Study IDs: 268347889
Record Dates: First submitted 2022-06-11; First posted 2022-06-15 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure; Self Care
Keywords: Heart Failure; Validity and Reliability; Self Care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Heart Failure Group — This is a single-center, prospective, observational study. The assessment and reporting will be followed the Consensus-Based Standards for the Selection of Health Status Measurement Instruments (COSMIN) checklist.
  Other Names: Assesment

SUMMARY:
The aim of this study was to evaluate the translation, cross-cultural fit, and psychometric properties of the European Heart Failure Self-Care Behavior Questionnaire for Caregivers.

DETAILED DESCRIPTION:
This research will be of descriptive type. The population of the study will be heart failure patients who applied to the University Hospital Cardiology clinic and polyclinic. The sample of the study will consist of patients who meet the research criteria and agree to participate in the study. The data collection tools of the study are the patient questionnaire (17 questions), the European Heart Failure Self-Care Behavior Scale for Caregivers (9 questions) and the Caregiver Contribution Scale in Heart Failure Self-Care, which was conducted by the researchers by scanning the literature.

English Turkish translations will be made before starting the research. Afterwards, expert opinion will be taken for the suitability of the scale items. Then, the Turkish scale items will be translated back into English and the linguist's opinion will be taken that the scale can be applied. Language and content validity will be done for the scale form. The scale items will be translated into Turkish and expert opinions will be taken. Then, the Turkish scale items will be translated back into English and the linguist's opinion will be taken that the scale can be applied. Language validity and content validity will be done in the study. Explanatory Factor Analysis will be applied for the validity of the questionnaire. Kaiser Meyer Olkin(KMO) Test, which measures the adequacy of sample size as antecedent tests, and Bartlett's Test For Sphericity will be used to test sphericity. Factor Analysis Principal Component Analysis Method will be applied.

ELIGIBILITY:
Inclusion Criteria:

* be over 18
* To be a caregiver for patients with heart failure for at least 1 year.
* Volunteer to participate in the research.

Exclusion Criteria:

* Having communication problems and mental problems.
* be under the age of 18.
* Receiving hemodialysis treatment for less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Heart Failure
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-06-12 (Actual); Primary Completion 2022-09-10 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
European Heart Failure Self-Care Behavior Scale for Caregivers | Baseline
  Using a five-point Likert scale, patients report the extent to which they agree with the statements corresponding to the 9-item self-care behavior (for example, weighing oneself every day), with responses ranging from "totally agree" to "disagree".
Scale of Caregiver Contribution in Heart Failure Self-Care | Baseline
  "Caregiver contribution scale in heart failure self-care", which consists of 22 items, consists of 3 separate scales.

CONTACTS AND LOCATIONS:
Overall Officials: İbrahim C Di̇ki̇ci̇, MSc, Study Director — Harran Üniversitesi
Locations (1):
- Harran University, Sanliurfa, Türki̇ye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No